CLINICAL TRIAL: NCT04423185
Title: Platform Study of Genotyping Guided Precision Medicine for Rare Tumors in China
Brief Title: PLATFORM Study of Precision Medicine for Rare Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ning Li, Chief, Office of Clinical Trial Center, CancerIHCAMS, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2380
Record Dates: First submitted 2020-05-27; First posted 2020-06-09 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Rare Tumor
Keywords: Rare tumor; NGS; actionable alterations; precision medicine; immunotherapy
MeSH Terms: interventions — aumolertinib; dacomitinib; alectinib; Crizotinib; pyrotinib; Imatinib Mesylate; niraparib; palbociclib; Vemurafenib; sintilimab; atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (17):
- Almonertinib-EGFR mutation (Experimental): Administration: 110 mg oral qd, to disease progression or intolerable adverse effects.
  Interventions: Drug: Almonertinib 110 MG
- Dacomitinib-EGFR mutation (Experimental): Administration: 45 mg oral qd, to disease progression or intolerable adverse effects.
  Interventions: Drug: Dacomitinib 45 MG
- Alectinib-ALK fusion (Experimental): Administration: 600 mg oral qd, to disease progression or intolerable adverse effects.
  Interventions: Drug: Alectinib 150 MG
- Crizotinib-ALK fusion (Experimental): Administration: 250 mg oral bid, to disease progression or intolerable adverse effects.
  Interventions: Drug: Crizotinib 250 MG
- Vemurafenib-BRAF mutation (Experimental): Administration: 960 mg oral bid, to disease progression or intolerable adverse effects.
  Interventions: Drug: Vemurafenib 240 MG
- Niraparib-BRCA mutation or HRD (Experimental): Administration: 200/300 mg oral qd, to disease progression or intolerable adverse effects.
  Interventions: Drug: Niraparib 200/300 MG
- Pyrotinib-HER-2 overexpression/amplification (Experimental): Administration: 400 mg oral qd, to disease progression or intolerable adverse effects.
  Interventions: Drug: Pyrotinib 160/80 MG
- Imatinib-CKIT mutation (Experimental): Administration: 400 mg oral qd, to disease progression or intolerable adverse effects.
  Interventions: Drug: Imatinib 400 MG
- Palbociclib-CDKN2A mutation (Experimental): Administration: 125 mg oral qd for 21 days q28d, to disease progression or intolerable adverse effects.
  Interventions: Drug: Palbociclib 125mg
- Crizotinib-ROS-1 fusion (Experimental): Administration: 250 mg oral bid, to disease progression or intolerable adverse effects.
  Interventions: Drug: Crizotinib 250 MG
- Crizotinib-C-MET amplification (Experimental): Administration: 250 mg oral bid, to disease progression or intolerable adverse effects.
  Interventions: Drug: Crizotinib 250 MG
- Crizotinib-C-MET mutation (Experimental): Administration: 250 mg oral bid, to disease progression or intolerable adverse effects.
  Interventions: Drug: Crizotinib 250 MG
- Pyrotinib-HER-2 mutation (Experimental): Administration: 400 mg oral qd, to disease progression or intolerable adverse effects.
  Interventions: Drug: Pyrotinib 160/80 MG
- Sintilimab-PD-1 (Experimental): Administration: 200mg q21d, to disease progression or intolerable adverse effects.
  Interventions: Drug: Sintilimab 100MG
- Combination ARM-Niraparib & Sintilimab (Experimental): Niraparib (200mg oral qd) combined with Sintilimab (200mg iv q21d) after acquired resistance to Niraparib.
  Interventions: Drug: Niraparib 200/300 MG; Drug: Sintilimab 100MG
- Combination ARM-Vemurafenib & Atezolizumab (Experimental): Vemurafenib (960 mg oral bid) & Atezolizumab (1200mg iv q21d) after acquired resistance to Vemurafenib.
  Interventions: Drug: Vemurafenib 240 MG; Drug: Atezolizumab 1680 MG
- Combination ARM-Palbociclib & Atezolizumab (Experimental): Palbociclib (125 mg oral qd for 21 days q28d) combined with Atezolizumab (1680mg iv q28d) after acquired resistance to Palbociclib.
  Interventions: Drug: Palbociclib 125mg; Drug: Atezolizumab 1680 MG

INTERVENTIONS:
Drug: Almonertinib 110 MG — Patients with advanced rare tumors who failed to standardized treatment carrying EGFR mutations will be administrated with Almonertinib.
  Other Names: HS-10296; AMEILE
  Arms: Almonertinib-EGFR mutation
Drug: Dacomitinib 45 MG — Patients with advanced rare tumors who failed to standardized treatment carrying EGFR mutations will be administrated with Dacomitinib.
  Other Names: Vizimpro
  Arms: Dacomitinib-EGFR mutation
Drug: Alectinib 150 MG — Patients with advanced rare tumors who failed to standardized treatment carrying ALK fusion will be administrated with Alectinib.
  Other Names: Alecensa
  Arms: Alectinib-ALK fusion
Drug: Crizotinib 250 MG — Patients with advanced rare tumors who failed to standardized treatment carrying ALK fusion, ROS-1 fusion, C-MET amplification, C-MET mutation will be administrated with Crizotinib.
  Other Names: Xalkori
  Arms: Crizotinib-ALK fusion; Crizotinib-C-MET amplification; Crizotinib-C-MET mutation; Crizotinib-ROS-1 fusion
Drug: Pyrotinib 160/80 MG — Patients with advanced rare tumors who failed to standardized treatment carrying HER-2 mutation or HER-2 over expression/amplification will be administrated with Pyrotinib.
  Other Names: SHR-1258
  Arms: Pyrotinib-HER-2 mutation; Pyrotinib-HER-2 overexpression/amplification
Drug: Imatinib 400 MG — Patients with advanced rare tumors who failed to standardized treatment carrying CKIT mutation will be administrated with Imatinib.
  Other Names: Gleevec
  Arms: Imatinib-CKIT mutation
Drug: Niraparib 200/300 MG — Patients with advanced rare tumors who failed to standardized treatment carrying BRCA1/2 mutation will be administrated with Olaparib.
  Other Names: Niraparix
  Arms: Combination ARM-Niraparib & Sintilimab; Niraparib-BRCA mutation or HRD
Drug: Palbociclib 125mg — Patients with advanced rare tumors who failed to standardized treatment carrying CDKN2A mutation will be administrated with palbociclib.
  Other Names: Ibrance
  Arms: Combination ARM-Palbociclib & Atezolizumab; Palbociclib-CDKN2A mutation
Drug: Vemurafenib 240 MG — Patients with advanced rare tumors who failed to standardized treatment carrying BRAF mutation will be administrated with Vemurafenib.
  Other Names: Zelboraf
  Arms: Combination ARM-Vemurafenib & Atezolizumab; Vemurafenib-BRAF mutation
Drug: Sintilimab 100MG — Patients with advanced rare tumors who failed to standardized treatment carrying no targeted alterations will be administrated with Sintilimab.
  Other Names: Tyvyt
  Arms: Combination ARM-Niraparib & Sintilimab; Sintilimab-PD-1
Drug: Atezolizumab 1680 MG — Patients with BRAF mutation treated with vemurafenib, after acquired resistance, will combine vemurafenib with atezolizumab.
  Other Names: TECENTRIQ
  Arms: Combination ARM-Palbociclib & Atezolizumab; Combination ARM-Vemurafenib & Atezolizumab

SUMMARY:
A Phase II, open label, non-randomized, multiple-arm, single-center clinical trial in patients with advanced rare solid tumors who failed to standard treatment.

DETAILED DESCRIPTION:
Based on the fact that a high incidence rate (14.2%) of rare tumor (incidence rate <2.5/100,000) as defined in this study according to the National Cancer Registry data from National Cancer Center of China, as well as the current status of lacking guidelines and consensus of rare tumor treatment. We proposed this study "A Phase II, open label, non-randomized, multiple-arm, single-center clinical trial in patients with advanced rare solid tumors who failed to standard treatment", aims to evaluate the safety and efficacy of targeted drugs of specific tumor-driven genes in patients with advanced rare solid tumors with corresponding actionable alterations, as well as the safety and efficacy of immune checkpoint (PD-1) inhibitors in patients with advanced rare solid tumors without actionable alterations. Patients with advanced rare tumors who failed to standardized treatment carrying actionable alterations as "EGFR mutation (exon 19 deletion mutation, L858R replacement mutation), ALK gene fusion, ROS-1 gene fusion, C-MET gene amplification or mutation (D1010 mutation, 14 exon mutation, y1003 mutation), BRAF mutation, CDKN2A mutation, BRCA1/2 mutation, HER-2 mutation, HER-2 over expression/amplification, C-KIT mutation", will enroll targeted therapy arms and be given corresponding targeted drugs (Dacomitinib, Crizotinib). And patients without targeted alterations mentioned above will enroll PD-1 inhibitor arm and to be treated with Sintilimab. After acquired resistance patients treated with olaparib and palbociclib will receive combination treatment with durvalumab. After acquired resistance patients treated with vemurafenib will receive combination treatment with atezolizumab. The statistics of current study adopts Simon's two-stage Minimax design: In the first stage of clinical research, 12 subjects will be observed. If the number of CR + PR is less than 1, the trial will be terminated, otherwise, the group will continue to expand to 16 subjects. Therefore, in the first stage, there are 12*5/(1-10%)=54 patients of targeted treatment group and 126 patients in the immunotherapy group, 180 patients totally in the first stage. If they all enter the second stage, the final target treatment group is 16*5/(1-10%) = 72 patients and the immunotherapy group which has 168 patients which brings to a total of 240 patients. The sample size of the study shall be adjusted according to the interim analysis. Primary Endpoint of this study is objective response rate (ORR) in immunotherapy group and targeted therapy group assessed by Blinded Independent Central Review (BICR) and investigator. Secondary Endpoints are Progression-Free Survival (PFS) in the targeted treatment group assessed by Blinded Independent Central Review and investigator; PFS (RECIST 1.1) and iPFS (iRECIST) in the single drug immunotherapy group assessed by Blinded Independent Central Review and investigator; Duration of Response (DoR) in the targeted therapy and single immunotherapy groups assessed by the investigator; Durable Clinical Benefit (DCB) in the single drug immunotherapy group; Incidence of Adverse Events (AE) in subjects ect.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, the age at the time of signing the informed consent is no less than 18 years old;
2. Patients with advanced or metastatic rare solid tumor confirmed by histological confirmed;
3. ECOG score is 0 or 1; ECOG score needs to be evaluated 7 days before the first treatment;
4. Expected survival ≥12 weeks;
5. According to Response Evaluation Criteria in Solid Tumor (RECIST 1.1), there is at least one imaging measurable lesions, which has obvious disease progress before radiotherapy or after radiotherapy;
6. Within the scope of CMPA approved drug indications, the disease has progressed after the standard treatment recommended by NCCN or CSCO guidelines (if there is standard treatment, the recommended level is IA-IIA), or there is no standard effective treatment plan, or it is no longer suitable for standard anti-tumor treatment, or the patients refuse the standard treatment plan;
7. Fresh biopsy tissue samples (obtained within 12 weeks before the first use of the drug, 4 pieces of coarse needle biopsy must be provided, and no other anti-tumor treatment, systemic anti infection treatment, vaccination, et al.) and peripheral blood samples must be provided for molecular typing;
8. Must have a primary or metastatic paraffin specimen (without radiotherapy) other than bone metastatic lesions before enrollment (within 2 years, 15-20 sheets, 4-6μm thick white slices, of which 5 need to be glued and baked ). If requirements are not met, investigator are allowed the decision to enroll subjects according to the specific situation.
9. If there is pleural or peritoneal effusion, the specimens must be taken for pathological cytological examination of which 300 ml samples must be provided;
10. In the condition that the primary lesions biopsy specimen has been provided, if the metastatic lesion is able to be biopsied, it is suggested to keep the specimen for pathological testing and provide fresh tissue specimen (optional); when obtaining EGFR mutation, ALK fusion, ROS-1 fusion, C-MET amplification, C-MET mutation, BRAF mutation, BRCA1/2 mutation, C-KIT mutation, HER-2 mutation HER-2 over expression/amplification, CDKN2A mutation patients will enroll in corresponding sub-study of targeted therapy; if no above mentioned actionable mutation is identified, patients will enroll immunotherapy sub-study. (Each sub-study has separate inclusion and exclusion criteria besides general ones)
11. After the progression of the subject's disease, if conditions permit, fresh tissue samples shall be obtained from the same biopsy lesions and the metastasis lesions of the previously obtained samples;
12. Toxic and side effects caused by previous treatment need to be restored to ≤ Grade 1 or returned to the baseline value (NCI-CTCAE version 5.0, except for hair loss);
13. Negative pregnancy test (only applicable for women with childbearing potential). No childbearing potential is defined as being postmenopausal for longer than one year or having undergone surgical sterilization or hysterectomy. All patients (male and female) agree to use an effective form of contraceptive measures and continue its use for the duration of treatment and within 8 weeks after the end of treatment;
14. Signed, written informed consent of volunteers that join the group shall follow the study treatment plan, follow-up plan and cooperate to observe the adverse events and efficacy.

Exclusion Criteria:

1. History of PD-1 / PD-L1 drug treatment.
2. History of the targeted drug treatment of this study.
3. Allergies towards drug ingredients or excipients in this study.
4. History of interstitial lung disease or radiation pneumonitis of any type.
5. Central Nervous System (CNS) metastases with brain metastases-related symptoms, which is not stable in neurology, or need to increase steroid dosage to control CNS disease. (Note: Patients with controlled CNS metastasis are eligible to participate in this study. Before entering the study, subject must have completed radiotherapy or CNS tumor metastasis surgery for more than fourteen days, neurological function must be in a stable state with no new neurological defects found in the clinical examination and no new problems found in the CNS imaging examination. If necessity arises for subjects to use steroids for CNS metastases treatment, said steroid treatment dose must have reached stable treatment for ≥ 3 months at least two weeks before entering the study.
6. Current uncontrollable third cavity effusion, such as a large amount of pleural effusion or ascites.
7. Unmeet the inclusion criteria of sub scheme.
8. Major surgical operations or incomplete healing of injury within 28 days prior to study treatment's first administration and chest radiotherapy of > 30 Gy within 6 months.
9. History of receiving other investigational drugs within 14 days or 5 half-lives (whichever is longer) prior to the first administration.
10. History of receiving live vaccine within 30 days prior to the first administration. Seasonal influenza vaccines that do not contain live viruses are allowed.
11. History of hypersensitivity to the active ingredients or non-active excipients of the study drug, hypersensitivity to drugs with chemical structure similar to the study drug or hypersensitivity to similar drugs of the study drug.
12. Current active infection requiring systemic treatment (antibiotics); or any of the following:

    1. HIV positive or known history of acquired immunodeficiency syndrome;
    2. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection is defined as HBsAg positive and the number of HBV DNA copies exceeds the upper limit of normal value, or HCV AB positive;
    3. Active tuberculosis (with exposure history or positive tuberculosis test; with clinical and / or imaging manifestations);
    4. Positive antibody of Treponema Pallidum.
13. Current evidenced uncontrollable systemic diseases (such as severe mental, neurological, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, liver or kidney diseases, uncontrolled hypertension [i.e., still greater than or equal to CTCAE Grade 3 hypertension after drug treatment]).
14. History of myocardial infarction, coronary artery / peripheral artery bypass or cerebrovascular accident within 3 months.
15. Diagnosed with a second type of malignant tumor within 5 years before the first diagnosis of a rare solid tumor (excluding completely resected basal cell carcinoma, bladder carcinoma in situ, cervical carcinoma in situ).
16. History of receiving of any organ transplantation, including allogeneic stem cell transplantation. Transplantation without immunosuppression (corneal transplantation, hair transplantation) is excluded.
17. Cardiovascular disease or symptom includes any of the following:

    1. History of Congestive Heart Failure requiring treatment and of New York Heart Association class III / IV CHF (see Appendix 3) ;
    2. Current ventricular arrhythmia requiring antiarrhythmic drugs treatment, or uncontrollable or unstable arrhythmia;
    3. Severe conduction disorder (such as grade II or III AV block);
    4. Angina requiring treatment;
    5. QT interval (QTC) of 12 lead ECG is ≥ 450 ms in male and ≥ 470 MS in female;
    6. History of congenital long QT syndrome, congenital short QT syndrome, torsade de pointe or pre-excitation syndrome;
    7. History of LVEF decline to below 50% determined by echocardiography or MUGA scan;
    8. History of myocardial infarction in the past 6 months.
18. Inadequate bone marrow reserve or organ function evidenced by the following laboratory results:

    1. Absolute value of neutrophils < 1.5 × 109 / L;
    2. Platelet count < 100 × 109 / L (transfusion dependent patients should be excluded from this study);
    3. Hemoglobin < 90g / L;
    4. ALT is > 2.5 x Upper Limit of Normal (ULN) If there is no clear liver metastases, ALT > 5 x ULN if there is liver metastases;
    5. Aspartate aminotransferase (AST) > 2.5 x ULN If there is no definite liver metastases. AST > 5x ULN if there is liver metastases;
    6. Total bilirubin > 1.5 x ULN if there is no liver metastases; Total bilirubin > 3 x ULN if there is definite Gilbert syndrome (Unconjugated Hyperbilirubinemia) or liver metastases;
    7. Creatinine > 1.5 x ULN with Creatinine clearance < 50 ml / min (measured value, or calculated value by Cockcroft Gault formula); Only when Creatinine > 1.5 x ULN, Creatinine clearance needs to be checked for confirmation;
    8. If bone metastasis is present and investigator concluded that liver function is adequate, the increase of ALP alone will not be excluded;
    9. Coagulation function: INR, PT, APTT> 1.5 times ULN (whether the patients using or not using anticoagulant drugs can be enrolled is determined by the investigator).
    10. Myocardial enzyme CK and CKMB test values are not in the normal range;
    11. The examination value of thyroid function is not within the normal range or it is not slightly abnormal but does not need treatment.
19. History of swallowing dysfunction, active gastrointestinal disease or other diseases that significantly affect the absorption, distribution, metabolism and excretion of oral drugs. The patients with history of subtotal gastrectomy. (Note: this standard is not applicable to the sub schemes with the investigational drug as injection).
20. Pregnant or lactating women.
21. Serious medical or mental illness that may affect program compliance and tolerance to treatment.
22. Those investigators believe that patients with other potential risks are not suitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Measured from first dose until confirmed response or progression, assessed up to 2 years.
  The percentage of patients with a confirmed Blinded Independent Central Review (BICR) and investigator-assessed complete or partial response according to Response Evaluation Criteria In Solid Tumours (RECIST) 1.1.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Measured from first dose until progression, assessed up to 2 years.
  The time from first dose until the date of objective disease progression or death (by any cause in the absence of progression).
iRECIST Evaluated Progression Free Survival (iPFS) | Measured from response until progression, assessed up to 2 years.
  The interval between the initiation of study treatment and the first documentation of CUPD (second confirmation of Disease Progression) or death due to any cause as defined by the iRECIST standard in the single drug immunotherapy group
Duration of Response (DoR) | Measured from response until progression, assessed up to 2 years.
  The time from the date of first response until date of disease progression or death in the absence of disease progression.
Disease Control Rate (DCR) | Measured from first dose until confirmed response or progression, whichever came first, assessed up to 2 years.
  The percentage of patients treated with targeted and single immunotherapy assessed by the investigator,
Durable Clinical Benefit (DCB) | Measured from first dose until confirmed response or progression, whichever came first, assessed up to 2 years.
  Partial Response (PR) or Complete Response (CR) or Stable Disease (SD) in the single drug immunotherapy group and without Disease Progression at more than six months.
Overall survival (OS) | Measured from first dose until death or final cohort data cut-off, whichever came first, assessed up to 2 years.
  The median survival time of patients
One year of Overall Survival rate (1-year OS rate) | Measured from first dose until death, assessed up to 2 years.
  Percentage of patients who is alive at 1-year from first dose of treatment.
Incidence of Adverse Events (AE) in subjects | Continuously from first dose to end of safety follow up after study treatment discontinuation, assessed up to 2 years.
  To evaluate safety and tolerability of each study treatment.
The 6-month PFS rate | Measured from response until progression, assessed up to 2 years.
  The proportion of patients who are alive and progression-free more than 6 months after the first dose of study therapy Progression-free Survival (PFS) the proportion of patients with PFS ≥ 6 months in the total enrollment since the start of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Doctor, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer hospital Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang S, Huang HY, Wu D, Fang H, Ying J, Bai Y, Yu Y, Fang Y, Jiang N, Sun C, Yu A, Fan Q, Xing S, Ni Y, Zhang W, Wu C, Ji X, Wang H, Guo Y, Tang Q, Wang Y, Tang Y, Li N. Platform study of genotyping-guided precision medicine for rare solid tumours: a study protocol for a phase II, non-randomised, 18-month, open-label, multiarm, single-centre clinical trial testing the safety and efficacy of multiple Chinese-approved targeted drugs and PD-1 inhibitors in the treatment of metastatic rare tumours. BMJ Open. 2021 Jun 3;11(6):e044543. doi: 10.1136/bmjopen-2020-044543. PMID 34083331